CLINICAL TRIAL: NCT00484094
Title: Post Marketing Surveillance Study To Observe Safety And Efficacy Of Rapamune
Brief Title: Study Investigating Rapamune For Post-Marketing Surveillance
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0468X1-4411; B1741015 (Other: Alias Study Number)
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Transplantation
Keywords: Rapamune; Safety; Efficacy; Kidney Transplantation
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rapamune
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — Dosage and treatment duration will be decided by physician's discretion considering patient's clinical situations
  Other Names: Rapamune

SUMMARY:
To provide safety and effectiveness information for Rapamune during the post-marketing period as required by Korea Food and Drug Administration (KFDA) regulations in order to identify any potential drug related treatment factors in the Korean population, such as:

1. Unknown adverse reactions, especially serious adverse reactions
2. To assess the incidence of adverse reactions under the routine drug uses
3. Factors that may affect the safety of the drug (e.g., proteinuria)
4. Factors that may affect the effectiveness of the drug

DETAILED DESCRIPTION:
All patients who receive Rapamune for certain period of time should be included as far as patients consent to participate

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 13 years or older receiving renal transplants, who are newly administered Rapamune after a contract is made between Pfizer Korea and an investigator and/or an institution for conducting this study.

Exclusion Criteria:

* Any patient who does not agree that Pfizer and companies working with Pfizer use his/her information.
* Patients who have known hypersensitivity to Rapamune or its derivatives or any excipients in the formulation.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who receive Rapamune after kidney transplantation
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2011-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- South Korea (11):
  - Seoul National University Hospital (SNUH), Seoul, Seoul
  - Yeungnam University Medical Center, Daegu
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Gyeonggi-do
  - Maryknoll Medical Center, Pusan
  - Kangdong Sacred Heart Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Korea University Anam Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Konkuk University Medical Center, Seoul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0468X1-4411&StudyName=Study%20Investigating%20Rapamune%20For%20Post-Marketing%20Surveillance

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between July 2011 and June 2015 from Korean health care centers.
Groups:
- Rapamune: Participants were administered Rapamune as part of routine practice. The use and dosage recommendations for Rapamune were based on the approved local product document and were adjusted solely according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Rapamune
Started | 209
Completed | 167
Not Completed | 42
Not completed — Discontinued | 39
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: Participants who received Rapamune at least once and were evaluated on its related safety endpoints at least once.
Arm/Group | Rapamune
Number analyzed (Participants) | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.93 (13.10)
Gender [Count of Participants; unit: Participants]
  Female | 81
  Male | 128
Type of Transplantation [Number; unit: Participants] — Primary transplantation: Participants received renal transplantation for the first time.
  Secondary transplantation: Participants received renal re-transplantation.
  Participants
    Primary Transplantation | 199
    Secondary Transplantation | 10
Type of Donation [Number; unit: Participants]
  Cadaveric | 76
  Living | 132
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)/Adverse Drug Reactions (ADRs), Serious AEs (SAEs)/Serious ADRs (SADRs), Unexpected AEs/ADRs, and Unexpected SAEs/SADRs
Description: All AEs reported after the start of administration of Rapamune were considered as treatment-emergent AEs and summarized. All AEs, except for those with causal relationship to the study drug assessed as "unlikely", were considered as AEs whose causal relationship to the study drug could not be excluded and classified as ADRs. Unexpected AEs/ADRs were classified by medical review with reference to the local product document and confirmed by Pfizer.
Time Frame: Six months (±1 month) after initiating Rapamune administration or until completion of Rapamune administration, whichever was earlier.
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Rapamune
Number analyzed (Participants) | 209
Percentage of participants
  AEs | 54.07
  ADRs | 43.06
  SAEs | 7.66
  SADRs | 2.87
  Unexpected SAEs | 2.39
  Unexpected SADRs | 0.48

2. Primary Outcome: Percentage of Participants With Clinically Significent Abnormal Laboratory Test
Description: Laboratory test was not mandatory because this study was a non-interventional study.
Time Frame: as for outcome 1
Population: This analysis was not performed because laboratory data were not collected during the study.
Arm/Group | Rapamune
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants With Biopsy-Confirmed Acute Rejection Using Banff 09 Diagnostic Categories for Renal Allograft Biopsies
Description: Renal biopsy was required to confirm the diagnosis of acute rejection. However, due to the non-interventional nature of this study, biopsy could not be mandatory. The decision of whether to perform a biopsy was made at the discretion of the investigator and the result was collected if performed.
Time Frame: At 6 months (±1 month) after initiating Rapamune administration or at the time of completion of Rapamune administration, whichever was earlier.
Population: Efficacy Analysis Set: Participants with efficacy data recorded on the case report form (CRF) at 6 months (±1 month) after initiating Rapamune administration or at the time of completing Rapamune administration (whichever was earlier) were included in the Efficacy Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rapamune
Number analyzed (Participants) | 209
Percentage of participants | 3.35 [0.91 to 5.79]

4. Secondary Outcome: Percentage of Participants Alive
Description: The investigator recorded the participant's survival status and evaluation date on the CRF.
Time Frame: as for outcome 3
Population: Efficacy Analysis Set; Participants who had available data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rapamune
Number analyzed (Participants) | 206
Percentage of participants | 99.51 [98.57 to 100.00]

5. Secondary Outcome: Percentage of Participants With Survived Graft
Description: Graft survival was defined as not showing graft loss at the time of evaluation.
Time Frame: as for outcome 3
Population: Efficacy Analysis Set; Participants who had available data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rapamune
Number analyzed (Participants) | 206
Percentage of participants | 99.51 [98.57 to 100.00]

6. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) Calculated by Nankivell Formula
Description: Graft function was evaluated by eGFR using Nankivell formula. The investigator recorded the date of evaluation and the calculated value on the CRF.
Time Frame: as for outcome 3
Population: Efficacy Analysis Set.
Measure: Median (Full Range); unit: mL/min
Arm/Group | Rapamune
Number analyzed (Participants) | 209
mL/min | 67.07 [4.80 to 113.27]

ADVERSE EVENTS:
Time Frame: Six months (±1 month) after initiating Rapamune administration or until completion of Rapamune administration, whichever was earlier.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Rapamune
Serious Adverse Events (participants affected / at risk) | 16/209
Other Adverse Events (participants affected / at risk) | 76/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rapamune (N=209)
Ascites (General disorders) | 1
Hypertension (Vascular disorders) | 1
Hyperparathyroidism (Endocrine disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Plasma osmolality increased (Metabolism and nutrition disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Angina pectoris aggravated (Cardiac disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Transplant rejection (Immune system disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Azotaemia (Renal and urinary disorders) | 4
Urinary tract disorder (Renal and urinary disorders) | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Polyomavirus infection (Infections and infestations) | 1
Abscess (Infections and infestations) | 1
Cystitis (Renal and urinary disorders) | 1
Infection susceptibility increased (General disorders) | 1
Herpes zoster (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rapamune (N=209)
Abdominal pain (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 10
Gastritis (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 7
Stomatitis ulcerative (Gastrointestinal disorders) | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 24
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 10
Urinary tract infection (Renal and urinary disorders) | 4
Coughing (Respiratory, thoracic and mediastinal disorders) | 3
Transplant rejection (Immune system disorders) | 4
Acne (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Azotaemia (Renal and urinary disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days